CLINICAL TRIAL: NCT06925191
Title: Assessment of Hamstring Flexibility, Static and Dynamic Core Muscles Endurance in Patients With Chronic Ankle Instability
Brief Title: Assessment of Torso Musculature and Hamstring Flexibility in Patients With Chronic Ankle Instability
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Ahmed Abdelaziz Saleh, principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005526
Record Dates: First submitted 2025-03-25; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: hamstring flexibility; 90-90 active knee extension; torso musculature

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Group A (Experimental): 29 affected ankles of both genders diagnosed with Chronic ankle instability (CAI) who met the inclusion criteria. Group B (Control): 29 matched non-affected with CAI — 1-90-90Active knee extension test 2.Core muscles endurance tests(a. The static endurance tests b. The dynamic endurance tests)
  Time Frame: 1 session

SUMMARY:
The purpose of this study is to assess torso musculature in terms of static and dynamic core muscle endurance tests and hamstring flexibility in non-athletic patients with unilateral chronic ankle instability.

DETAILED DESCRIPTION:
Ankle sprains are extremely common in public as well as in sports. Most people with acute ankle sprains respond well to conservative treatment , but many may experience chronic ankle pain and instability .

Injuries to the ankle lateral ligament typically occur when the ankle joint is inverted and plantar flexed . Ankle sprains occur about seven times per 1000 person-years in the general population, and in highly active people, the incidence can reach 45 times per 1000 person-years .

Chronic ankle instability (CAI), which includes both functional and mechanical ankle instability, is characterized by recurrent ankle sprains, persistent symptoms, and a tendency to "giving way" .

The terms mechanical ankle instability (MAI) and functional ankle instability (FAI) refer to two different conditions: FAI is defined as recurrent ankle sprains or re-damage, while MAI is defined as a state of ligament relaxation detected by objective physical examinations of the talar tilt and anterior drawer sign. The complaint of subjective feelings, such as ankle giving away in FI, is associated with FAI .

In relation to postural stability, which is characterized as the capacity to sustain and regulate one's center of gravity over a support base, postural control is a complicated process that arises from the cooperation and synergy of the vestibular, ocular, and somatosensory systems. Moreover, lower limb injuries are thought to be associated with postural instability.

In the kinetic chain that runs from the foot to the lumbar spine, core stability has been emphasized as a crucial factor to keep in mind when preserving dynamic joint stability .

It is important to note that in this instance, core stability refers to the hip complex's ability to maintain homeostasis following a disturbance and to avoid buckling. Additionally, there is clear evidence linking lower limb movement to trunk muscle activity . Motor chain disruptions resulting from dysfunction in the trunk, pelvis, and hips can cause lower extremity injuries and lower back pain (LBP) .

Additionally, the torso musculature was measured by testing the endurance of the core muscles (static and dynamic). The Bench Trunk Curl-Up test (BTCT) was used to measure dynamic endurance, while the modified right side-bridge, modified left side-bridge, trunk flexion and horizontal back extension tests were used for static endurance (the endurance time of each isometric test was recorded).

In addition to disorders including low back discomfort and irregular gait, tight hamstrings are linked to dysfunction in the lumbar spine, pelvis, and lower limb .

Tight hamstrings are linked to poor motor control patterns, which compromise postural muscle activation and make the hamstrings function more as stabilizers than as main movers. Hamstring tightness manifests because of this basic change in function .

Numerous research has assessed CAI's proximal deficiencies. A few evaluated their strength , and excitability Moreover, alterations in kinematics have been evaluated .

Statement of the problem

This study will try to answer the following question:

Are torso musculature and hamstring flexibility affected in non-athletic patients with unilateral chronic ankle instability? Purpose of the study The purpose of this study is to assess torso musculature in terms of static and dynamic core muscle endurance tests and hamstring flexibility in non-athletic patients with unilateral chronic ankle instability.

Hypotheses

It will be hypothesized that:

1. There is no significant difference in torso musculature in terms of static core muscle endurance between non-athletic healthy participants and non-athletic patients with unilateral chronic ankle instability.
2. There is no significant difference in torso musculature in terms of dynamic core muscle endurance between healthy participants and non-athletic patients with unilateral chronic ankle instability.
3. There is no significant difference in hamstring flexibility between non-athletic healthy participants and non-athletic patients with unilateral chronic ankle instability.

Significance of study Lateral ankle sprain is one of the most common sports injuries, and it has the highest recurrence rate among all lower-extremity musculoskeletal injuries .

chronic ankle instability (CAI) is linked to a lower lifetime quality of life, a lower degree of physical activity, and a higher chance of developing osteoarthritis in the joints .

Ankle sprains occurred 3.29 times per 1000 people annually in US emergency rooms in 2010 . The prevalence of CAI after a sprain is 25% overall, and in otherwise healthy adolescent athletes, it is 20% after an ankle sprain, even though over 15% of cases result in CAI, the public still views ankle sprains as benign injuries .

Hip muscle abnormalities are becoming more common in CAI patients, as described in studies , which might worsen the condition by impairing trunk and pelvic stability and causing the lower body to be malposition as a result .

Reduced lumbopelvic stability may theoretically exacerbate CAI, however this association is still theoretical. Tests that test a person's capacity to maintain hip and trunk alignment can be used to assess lumbar stability. However, no research has up to this point compared to the performance levels of those with and without CAI. Additionally, muscle deficiencies in the hip and trunk can impact lumbopelvic stability. There is, however, a lack of data on the anatomy of the trunk muscles in patients with CAI .

According to previous research, those with CAI experience higher rates of low back pain , delayed trunk muscle activation.

Previous study has investigated the relationship between core stability (CS) and CAI and concluded that, the lack of a clear correlation between trunk endurance and CAI remains unclear; nevertheless, it's possible that the McGill core endurance tests don't accurately assess lumbo-pelvic stability in CAI patients or distinguish between those who have the condition from those who don't. The individuals' sensorimotor systems were not sufficiently challenged by the tests to identify variations between groups. These tests only evaluate the static core endurance.

Therefore, it is crucial to assess torso musculature with CAI for both genders by both static and dynamic core endurance as This facilitates prevention of injury and management of the associated musculoskeletal deficits of CAI.

Previous research evaluating the Arthrogenic Muscle Response of the Hamstrings and Quadriceps with Chronic Ankle Instability produced the conclusion that participants with unilateral CAI had ipsilateral facilitation of the quadriceps and bilateral arthrogenic inhibition of the hamstrings. The motoneuron pool excitability in muscles acting on joints proximal to the ankle seems to be changed in individuals with unilateral CAI. Furthermore, deficiencies in sagittal plane force production were noted at the ankle and the knee, even though the source of instability was at the ankle.

The knee flexor muscles' maximal and submaximal isometric strengths as well as the knee extensor muscles' submaximal strengths are abnormal in people with CAI.

Previous studies assessed hamstring flexibility in ankle sprain or CAI in order to orient the therapist to evaluate the proximal affection that far from the injured site that influencing both preventative and therapeutic approaches to patient care, subsequently completing the evaluation procedures, reduce recurrence rate, restore functional loss and prevent degenerative sequels and concluded that CAI subjects have proximal muscular affection include hamstring tightness which may alter sacroiliac joint stability and subsequently back pain .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria was based on the standard criteria outlined by the International Ankle Consortium (Gribble et al., 2014).

  1. Their ages range from 20- 35 years old including both genders (male & female).
  2. Their BMI was 18.5- 30 kg/m2.
  3. A history of the previously injured ankle joint "giving way," and/or recurrent sprain, and/or "feelings of instability."
  4. Report episodes of giving way and sense of instability of the affected ankle
  5. Cumberland Ankle Instability Tool (CAIT) patient scores < 24.

Exclusion Criteria:

* Subjects were excluded if they have any of the following criteria:( Gribble et al., 2014).

  1. A history of previous surgeries on the musculoskeletal structures (i.e., bones, joint structures, nerves) in either lower extremity.
  2. A history of a fracture in either lower extremity requiring realignment.
  3. Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months that impacted joint integrity and function (i.e., sprains, fractures), resulting in at least 1 interrupted day of desired physical activity.
  4. Any patient received physical therapy treatment or medical treatment (NSAID)in the last 2weeks Before enrollment in the study.
  5. Any patients suffered from low back pain, lumbar disorder and Sacro iliac joint pain.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 29 healthy people and 29 non-healthy people with chronic ankle instability
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
90-90Active knee extension test | 1 session
  The angle of knee extension was measured in degrees by a standard goniometer while the patient in supine position and the hip was in 90 degrees of hip flexion

SECONDARY OUTCOMES:
Static Core muscles endurance tests | 1 session
  1. Modified Right side-bridge test was measured in second by stopwatch while the patient was told to lie on her right side with their right hip and elbow (which were flexed to a 90-degree angle) supporting their right side and their hips were elevated off the table.
  2. (Modified Left side-bridge test) The same procedures were repeated but for the left side
  3. Trunk flexors endurance test was measured in second by stopwatch while the patient was instructed to place her body against a wedge at a neutral head position, 90° hip and knee flexion, and 60° trunk flexion to begin the test. Each person had their arms folded across their chests. The examiner then shifted the wedge aside and gave the subject instructions to maintain her posture without using her back support
  4. Modified Biering-Sorensen test was measured in second by stopwatch while the patient was in prone position, supporting their lower legs on the table while maintaining their trunk straight out of the table .

OTHER OUTCOMES:
Dynamic Core muscles endurance test | 1 session
  Bench Trunk Curl-Up test was measured as how many repetitions was done in two minutes by stopwatch while The subject laid supine on a bench with their hips and knees bent to a 90-degree angle (using an extendable goniometer). The hands held the elbow on the other side of the crossed arms. Completed a trunk flexion, or "curl-up," until their elbows contact their thighs, their scapulae remain off the mat, and their heads neutral. They then go back to their starting positions.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt